CLINICAL TRIAL: NCT06139510
Title: Predictors of Pain Severity and Pain-Related Outcomes in Individuals With Sickle Cell Disease
Brief Title: Predictors of Pain in Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00112024; 1K01HL169339-01 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease; Chronic Pain
Keywords: quantitative sensory testing; pain sensitization
MeSH Terms: conditions — Anemia, Sickle Cell; Chronic Pain

STUDY DESIGN:
Masking Description: This study does not involve drug or biologic products. Masking is non-applicable.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals living with sickle cell disease (Other): Participants living with sickle cell disease will undergo standardized testing called quantitative sensory testing. Quantitative sensory testing measures changes in sensitivity to different type of sensations that include temperature, touch or pressure.
  Interventions: Other: Quantitative sensory testing

INTERVENTIONS:
Other: Quantitative sensory testing — Quantitative sensory testing is a standard type of pain testing that measures changes in sensitivity to different type of sensations that include temperature, touch or pressure.

SUMMARY:
Sickle cell disease is a painful inherited disorder that affects approximately 100,000 people in the United States, and more than half of these individuals develop chronic or persistent pain that is often severe and disabling. The factors that predict whether an individual with sickle cell disease will develop severe, disabling pain are unclear. The goal of this project is to identify the factors that predict severe pain outcomes in individuals living with sickle cell disease in order to improve pain management strategies and guide future studies of non-opioid therapies for treatment of their pain.

Participants who agree to enroll in this study will be asked to participate in a virtual and then an in-person study visit for their full initial study assessment. They will answer survey questions during the virtual visit, and will be asked to complete several types of standard testing to understand how their body handles pain during the in-person visit. After completing the virtual and in-person sessions, participants will receive text or electronic medical record messages with brief survey (will take less than 8 minutes to complete) on their pain experiences every three months until the study is completed (or up to 48 months for people who are enrolled at the beginning of the study).

DETAILED DESCRIPTION:
Severe, disabling pain is the hallmark of sickle cell disease (SCD). SCD pain is associated with poor quality of life, early mortality, and high healthcare costs. Clinicians face great challenges in managing SCD pain because of the poor understanding of the etiology of chronic/persistent SCD pain and the absence of validated clinical predictive tools that can accurately identify individuals with SCD who are at risk of developing severe, persistent pain with associated physical and/or psychological disability. The overall objective of this study is to identify predictors of pain severity and pain-related outcomes in SCD using a prospective, longitudinal study design. This proposal is supported by the hypothesis that pain-specific psychological and sensory factors are strong, modifiable predictors of SCD pain severity and pain-related outcomes. The understanding of pain-specific psychological and sensory predictors of SCD pain outcomes is anticipated to have important implications for (1) identifying SCD patients who are at risk for severe pain outcomes, (2) informing preventive and therapeutic management of SCD pain, and (3) selecting patients for clinical trials of non-opioid interventions for SCD pain. The hypothesis will be tested by pursuing two specific aims: Aim 1) Determine psychological predictors of pain outcomes; and Aim 2) Ascertain the strength of pain distribution and sensitivity as predictors of pain outcomes. The researchers will use reliable and well validated pain-specific patient-reported outcome (PRO) questionnaires to evaluate the strength of psychological factors for predicting pain severity and other pain-related outcomes in the study cohort (Aim 1) and will use body mapping and quantitative sensory testing (QST) to examine sensory predictors of pain outcomes (Aim 2).

ELIGIBILITY:
All participants must be between 15 and 40 years old and must be able to provide informed, written consent (for adults) or parental consent (for participants younger than 18 years).

Inclusion Criteria:

1. Diagnosis of sickle cell disease (documentation of SS, SC, S beta + thalassemia, S beta + thalassemia) is required
2. Participants must have had at least one sickle cell related pain episode that required treatment with opioids at home or in the hospital 12 months prior to recruitment
3. Participants who are on chronic analgesics (NSAID, acetaminophen) or opioids should be on a stable dose for 4 weeks prior to recruitment.

Exclusion Criteria:

1. Age less than 15 or greater than 40 years
2. Participants lacking the cognitive or mental capacity to assent to and complete study procedures
3. Pregnant females
4. Participants with history of a stroke with ongoing physical impairment that prevents participation in study procedures.
5. Participants with history of severe vaso-occlusive pain crisis resulting in either evaluation in an emergency department or admission to a hospital two weeks prior to study enrollment.
6. Current or active infection
7. Any condition that the principle investigator considers would preclude or bias participation in the study, such as (1) neuropathy from diabetes or other causes, (2) active avascular necrosis requiring treatment for pain

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain pain severity | At baseline and every three months while enrolled in the study, up to 48 months
  Will be determined by answering the severity subscale of the Brief Pain Inventory

SECONDARY OUTCOMES:
Change in psychological distress | At baseline and every three months while enrolled in the study, up to 48 months
  Will be determined based on answers to the anxiety and depression subscales of the PROMIS-29 questionnaire. A composite score of the subscales will be reported.
Change in pain interference | At baseline and every three months while enrolled in the study, up to 48 months
  Will be determined based on answers to the pain interference subscale of the PROMIS-29 questionnaire.
Change in physical function | At baseline and every three months while enrolled in the study, up to 48 months
  Will be determined based on answers to the physical function subscale of the PROMIS-29 questionnaire.
Change in healthcare utilization for pain | At baseline and every three months while enrolled in the study, up to 48 months
  Will be determined based on answers to the PhenX Frequency of Sickle Cell Pain Episodes Per year questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Kenney, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No